CLINICAL TRIAL: NCT01860482
Title: An 8-weeks, Multicenter, Single Arm, Non-comparative, Phase 4 Clinical Trial to Assess the Efficacy and Safety of Newrabell® Tab. at 10mg b.i.d in Patients With Refractory Reflux Esophagitis(rGERD) to the Prior Standard PPIs Regimen
Brief Title: The Study to Evaluate Efficacy and Safety of Newrabell® Tab.(Rabeprazole Sodium) 10mg b.i.d in Refractory GERD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243GERD13003
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Reflux Esophagitis
Keywords: Refractory Reflux Esophagitis; GERD; Phase 4
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Newrabell single arm (Experimental): Newrabell® Tablet 10mg b.i.d PO during 8 weeks
  Interventions: Drug: Newrabell® Tablet 10mg

INTERVENTIONS:
Drug: Newrabell® Tablet 10mg
  Other Names: Rabeprazole sodium

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Newrabell® Tab. in patients with refractory reflux esophagitis to the prior standard PPIs regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged ≥ 20 years
2. Reflux esophagitis with erosion or ulceration confirmed by endoscopic exam.
3. Refractory reflux esophagitis to PPIs standard treatment as follows

   1. Ongoing heartburn symptom with or without these GERD-related symptoms : Regurgitation, Non-cardiac chest pain, Epigastric pain, Belching, Bloating, Satiety, Sore throat, Cough, Laryngitis, Hoarseness, Nausea, Vomiting, Dysphagia, Odynophagia, Weight loss
   2. Ongoing heartburn symptom with or without erosion ≥ grade A according to LA Classification
4. Ongoing heartburn symptoms ≥ 2 days during 1week right before administering first dose of IP
5. Decided to participate and signed on an informed consent form willingly

Exclusion Criteria:

1. Existence of upper gastrointestinal bleeding or active gastroduodenal ulcer at screening
2. History of operation in esophagus, stomach or duodenum
3. The following medical history

   1. Primary esophageal motility disease, Achalasia, Scleroderma, Esophageal/pyloric stricture, Primary esophageal spasm
   2. Barrett's esophagus ≥ 3 cm
   3. Zollinger-Ellison syndrome
   4. Infectious or inflammatory bowel disease, Severe malabsorption
4. Severe chronic heart failure, cardiovascular disease, renal failure, COPD, asthma, liver cirrhosis
5. History of cancer within 5 years, except completely recovered skin cancer
6. ALT or AST ≥ Upper limit of normal range X 3
7. Need antibiotics due to severe infection
8. Severe medical disease that needs these prohibited medication

   * Anticoagulant(Heparin, Warfarin, etc.), High dose of aspirin(>325mg/d), Digitalis(Digoxin, etc.), Diuretics, Atazanavir, NSAIDs or Steroids
9. Use PPIs or H2RA medicine within 1 week before administering first dose of IP, or need other PPIs or H2RA medicine during trial period
10. Allergy or hypersensitivity to IP or similar chemical structure(Benzimidazol derivatives, etc.)
11. Pregnant or breast-feeding women
12. Conversation impairment because of alcohol, drug addiction or mental illness, etc.
13. Administration of other IP within 28 days
14. Inability to record heartburn diary card
15. In investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Time to onset of first 1Day Heartburn free, Days | up to 8 weeks

SECONDARY OUTCOMES:
Time to onset of first 2Days Heartburn free, Days | up to 8 weeks
1Day Heartburn free days, % | up to 8 weeks
Time in Daytime of first Heartburn free, Days | up to 8 weeks
Time in Nighttime of first Heartburn free, Days | up to 8 weeks
Weekly Heartburn Improvement Rate, % | up to 8 weeks
Average Daytime and Nighttime Heartburn Score Change at W4 | up to 8 weeks
Average Daytime and Nighttime Heartburn Score Change at W8 | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jongsun Rew, Ph.D, Principal Investigator — Chonnam National University Hospital; Sungbum Cho, Ph.D, Principal Investigator — Chonnam National University Hospital
Locations (2):
- South Korea (2):
  - Chonnam National University Hospital, Gwangju, Donggu, Jebongro
  - Chonnam National University Hwasun Hospital, Gwangju, Hwasun-eup,Hwasun-gun